CLINICAL TRIAL: NCT03943303
Title: Effect of Monazite Sands in Patients With Osteoarthritis of the Knee
Brief Title: Effects of Sand Treatment on Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because the Pandemia COVID-19 was not possible to bring the participants to the beach.
Sponsor: University Vila Velha (Other)
Responsible Party: Principal Investigator, Denise Coutinho Endringer, Director of Research and graduate program, University Vila Velha
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: T015-M02-2019AF002; TO#617/2018 (Other Grant/Funding Number: FUNCITEC/MCI)
Record Dates: First submitted 2019-04-29; First posted 2019-05-09 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Osteo Arthritis Knee
Keywords: monazitc sands; radiation

STUDY DESIGN:
Intervention Model Description: The study will be carried out on the beaches of Areia Preta de Guarapari (source of monazitic sands) and on the beach of Itapoã in Vila Velha (sand without radiation). Selected patients will have their knees fully covered with beach sand, properly analyzed for radioactivity and temperature, for 30 minutes on 2 mornings a week for a period of 1 (one) year.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is unaware of the treatment that the patients received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural gamma radiation from the monazite sands (Experimental): Patients selected for the study will have their knee (s) affected by osteoarthrose fully submerged in the monazite beach sand 2 (two) times per week for 30 (thirty) minutes each session at the same location and at the same time of day. The natural gamma radiation doses of the monazite sands will be monitored, the radiation measurements gamma will be associated with the atmospheric and climatic measurements of each group. It is understood here as atmospheric measurements, level of solar radiation, spectrum of sunlight at the time of exposure, humidity, wind speed, ultraviolet radiation level, amount of ions present in the air and measurements of the magnetic field in the place.
  Interventions: Radiation: Natural gamma radiation from the monazite sands
- Normal sands exposure patients (Placebo Comparator): Patients selected for the study will have their knee (s) affected by osteoarthrose fully submerged in the no-monazite beach sand 2 (two) times per week for 30 (thirty) minutes each session at the same location and at the same time of day. To ensure the absence of radiation, mesuaraments of possible radiation will be monitored.
  Interventions: Radiation: Normal sands exposure patients

INTERVENTIONS:
Radiation: Natural gamma radiation from the monazite sands — Patients selected for the study will have their knee (s) affected by osteoarthrose fully submerged in the monazite beach sand 2 (two) times per week for 30 (thirty) minutes each session at the same location and at the same time of day.
  Other Names: Natural beach black sands
  Arms: Natural gamma radiation from the monazite sands
Radiation: Normal sands exposure patients — Patients selected for the study will have their knee (s) affected by osteoarthrose fully submerged in the no-monazite beach sand 2 (two) times per week for 30 (thirty) minutes each session at the same location and at the same time of day.
  Other Names: No-monazite sands
  Arms: Normal sands exposure patients

SUMMARY:
2528/5000 Historically the city of Guarapari / ES is known as the city health by the popular therapeutic effect of its sands in diverse diseases. The articular diseases are among the list of the aggravations that popularly the monazitic sands exert some therapeutic effect, emphasizing. Rheumatic diseases include osteoarthritis of the knee. It is a disease with a high prevalence and in recent years have presented an increase in the incidence supposedly caused by the aging population and due to the epidemic of obesity. Osteoarthrosis is proven to be a disease that leads to the incapacity and restriction of the individual's ability to come and go with high monetary costs for the patient and the government. In view of these facts presented, the objective is to investigate the therapeutic potential of monazite sands in elderly patients submitted to serial, controlled and standardized exposure, compared to patients exposed to beach sand without radiation.

DETAILED DESCRIPTION:
A sample of 150 patients with primary knee osteoarthrosis will be selected for the study, divided into two random groups that will be exposed to sand (one monazite sand group and another beach sand group without radiation) for 12 months. The groups will be evaluated at time 0 (at the patient's arrival in the group) and at 1, 2, 3, 6, 9 and 12 months of exposure following the literature criteria for evaluation of knee osteoarthrosis (Visual Analogue Scale (EVA) and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)) and non-specific and specific biomarkers (C-reactive protein, erythrocyte sedimentation rate, IL-1β, IL-6, IL-8, TGF-β, and TNF-α). In addition, the groups will undergo an initial interview and monitoring of the pharmacological therapies used prior to the study and during the months of follow-up using the Dáder methodology of pharmaceutical care adapted to the study. As a result, the scientific evidence of the efficacy of monazitic sands in knee osteoarthrosis is expected not only by clinical criteria but also by laboratory evidence on the markers of the inflammatory and degenerative process that allow us to document the real value of the monazitic sands for health of the population, to establish a great line of research for the state of Espírito Santo and to value the State of Espírito Santo and the municipality of Guarapari as potential itineraries for SPA tourism (aiming to improve health).

ELIGIBILITY:
Inclusion Criteria:

* Joint pain related to daily activities;
* No morning joint stiffness greater than 30 minutes;
* Age between 30 and 95 years.

Exclusion Criteria:

* History of previous knee surgery.
* History of fracture in the knee region.
* History of any secondary OA associated with any cystic arthropathy.
* Any treatment for the knee with methotrexate.
* History of hemorrhagic disorders.
* History of any infiltration of the knee during the previous 6 months (eg corticosteroids and hyaluronic acid).
* Morbid obesity.
* History of severe psychiatric disorders.
* History of skin cancer.

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Change in the Visual analgesic scale (0-10) | 1, 3, 6, 8 and 12 months
  Change pain perception through the visual analgesic scale of the volunteers. It consists of a graduated scale of 0 to 10 with regular intervals where zero means absence of pain and 10 is the maximum pain already experienced by the patient.

SECONDARY OUTCOMES:
Change total score (0 - 96) the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)- (lower scores indicate lower levels of symptoms or physical disability) | 1, 3, 6, 8 and 12 months
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire comprises three subscale. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.
Change the number of patient with higher concentration of Nonspecific inflammatory markers | 1, 3, 6, 8 and 12 months
  Quantification of nonspecific inflammatory markers (HSV and CRP) and specific (IL-1β, IL-6, IL-8, IL-17, TNF-α and TGF-β) per patient
Change the frequency of Self-medicatition to treat pain | 1, 3, 6, 8 and 12 months
  Evaluation of the frequency of self-medication before and during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: DENISE C Endringer, Dr, Principal Investigator — UVila Velha
Locations (1):
- Denise Coutinho Endringer, Vila Velha, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510
- [Result] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- See also: The Global Health Network template. — http://www.theglobalhealthnetwork.org

DOCUMENTS (8):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Protocol and statistical analysis (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03943303/Prot_SAP_ICF_000.pdf
  • Study Protocol and Informed Consent Form: Inform consent (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03943303/Prot_ICF_001.pdf
  • Study Protocol: Pharmaceutical care (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT03943303/Prot_002.pdf
  • Study Protocol: Screening_log (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT03943303/Prot_003.pdf
  • Study Protocol: Enrolment _log (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03943303/Prot_004.pdf
  • Study Protocol: Withdrawal_log (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT03943303/Prot_005.pdf
  • Study Protocol: Telephone_Contact_Log (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT03943303/Prot_006.pdf
  • Study Protocol: Meeting_minutes_template (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03943303/Prot_007.pdf